CLINICAL TRIAL: NCT03127020
Title: Open-Label, Non-Randomized Phase 2 Study With Safety Run-in Evaluating Efficacy and Safety of PQR309 in Patients With Relapsed or Refractory Lymphoma
Brief Title: Phase 2 Study With PQR309 in Relapsed or Refractory Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PIQUR Therapeutics AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other); University Hospital Munich (Other); University Hospital Freiburg (Other); Charite University, Berlin, Germany (Other); University of Stuttgart (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQR309-002A
Record Dates: First submitted 2016-04-14; First posted 2017-04-25 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Phosphatidylinositol 3-Kinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PQR309 (Experimental): PQR309 being taken continuously on daily basis (60,80mg) or intermittent (120mg, 140mg, 160mg) dosing
  Interventions: Drug: PQR309

INTERVENTIONS:
Drug: PQR309 — taken continuously on daily basis (60mg, 80mg) or intermittent dosing (120mg, 140mg, 160mg)
  Other Names: PI3K Inhibitor (phosphatidylinositol 3-kinase)

SUMMARY:
The main goal of this study is to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D) as well as preliminary antitumor activity of PQR309 administered orally, as once daily capsules continuously and on intermittent schedule, in patients with relapsed or refractory lymphomas.

DETAILED DESCRIPTION:
Open-label, non-randomized, multicentre phase 2 study with a safety run-in evaluating efficacy and safety of PQR309 in patients with relapsed or refractory lymphoma.

The maximum tolerated dose (MTD) of PQR309 in patients with advanced solid tumours was defined as 80 mg once daily given continuously (q.d. schedule) in a previous phase 1 study [8]. The safety run-in of this study will follow a modified 3 + 3 design to evaluate the safety of 60 and 80 mg PQR309 in patients with relapsed or refractory lymphoma administered p.o. once daily during a DLT (dose-limiting toxicity) period of 28 days.

In the safety run-in, three patients will be treated at 60 mg PQR309 for 28 days. Enrollment and treatment of all three patients may occur simultaneously as 80 mg PQR309 p.o. qd was established as the MTD maximum tolerated dose in solid tumours. Unless a DLT (dose-limiting toxicity) is observed in any of the three patients during the first 28 days of treatment, the investigators and the sponsor will decide to escalate the dose to 80 mg.Intermittent dosing schedules may be evaluated if, based on the overall evaluation of all the clinical and PK (pharmacokinetic) data from this and other studies with PQR309, data emerge during the step 1 of the phase 2 expansion in this PQR309 002A study, indicating that daily dosing of PQR309 is not adequately tolerated or inefficacious.

Intermittent dosing schedules may be evaluated if, based on the overall evaluation of all the clinical and PK (pharmacokinetic) data from this and other studies with PQR309, data emerge during the step 1 of the phase 2 expansion in this PQR309 002A study, indicating that daily dosing of PQR309 is not adequately tolerated or inefficacious.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed diagnosis* of relapsed or refractory lymphoma, received at least two prior lines of therapy regardless of transformation status. Patients with relapsed chronic lymphoid leukemia (CLL) are eligible if they have received one or more prior lines of any approved standard therapy * archival biopsies may be used if obtained up to a year prior to enrollment; re-biopsy is strongly recommended if last biopsy was obtained more than a year ago.
2. Only for patients in the Phase 2 part: At least one measurable nodal or extra-nodal lesion defined as follows: Clearly measurable (i.e. well-defined boundaries) in at least two perpendicular dimensions on imaging scan with > 1.5 cm in longest transverse diameter.
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1 (See Appendix 2).
5. Adequate organ system functions defined as:

   1. Absolute neutrophil count (ANC) ≥1.0x109/l
   2. Platelets ≥ 75x109/l
   3. Haemoglobin ≥ 85g/L
   4. Adequate hepatic function, defined as total bilirubin ≤ 1.5 times the upper limit of normal (ULN) and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN
   5. Adequate renal function, defined as serum creatinine ≤ 1.5 times ULN
   6. Fasting glucose < 7.0 mmol/L
6. Ability and willingness to swallow and retain oral medication.
7. Willingness and ability to comply with the trial procedures
8. Female and male patients with reproductive potential must agree to use effective contraception from screening until 90 days after discontinuation of PQR309
9. Signed informed consent1.5 cm in longest transverse diameter.

3. Age >18 years 4. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-1 5. Adequate organ system functions defined as:

1. Absolute neutrophil count (ANC) >1.0x109/l
2. Platelets > 75x109/l

Exclusion Criteria:

Any of the following conditions precludes enrollment of a patient:

1. Immunosuppression due to:

   * Allogeneic hematopoietic stem cell transplant (HSCT)
   * Any immune-suppressive therapy within 4 weeks prior to trial treatment start
2. Autologous stem cell transplant within 3 months prior to trial treatment start.
3. Concomitant anticancer therapy (e.g. chemotherapy, radiotherapy, hormonal therapy, immunotherapy, biological response modifier, signal transduction inhibitors and steroids (steroids as maintenance for adrenal insufficiency are allowed)).
4. Concomitant treatment with medicinal products that increase the pH (reduce acidity) of the upper gastrointestinal tract, including, but not limited to, proton-pump inhibitors (e.g. omeprazole), H2-antagonists (e.g. ranitidine) and antacids. Patients may be enrolled in the study after a wash-out period sufficient to terminate their effect (section 11.1.3.7).
5. Use of any investigational drug within 21 days prior to trial treatment start.
6. Patients who experienced National Cancer Institute (NCI) Common Terminology Criteria For Adverse Events (CTCAE) grade 4 on PI3K/mTOR inhibitors
7. Any major surgery, chemotherapy or immunotherapy within 21 days prior to trial treatment start.
8. Symptomatic or progressing central nervous system (CNS) involvement. Exception: Patients with meningeal involvement can be included upon discussion between the sponsor and the investigator.
9. Persisting toxicities NCI CTCAE ≥2 related to prior anticancer therapy
10. Presence of gastrointestinal disease or any other condition that could interfere significantly with the absorption of the study drug.
11. Severe/unstable angina, myocardial infarction or coronary artery bypass within the last 3 years prior to trial treatment start, symptomatic congestive heart failure New York Heart Association (NYHA) Class 3 or 4, hypertension BP>150/100mmHg
12. A serious active infection (e.g. chronic active hepatitis) at the time of treatment, or another serious underlying medical condition that could impair the ability of the patient to receive treatment.
13. Lack of appropriate contraceptive measures (male and female)
14. Pregnant or lactating women
15. Known HIV infection
16. Significant medical conditions which could jeopardize compliance with the protocol.
17. Uncontrolled diabetes mellitus; patients with controlled diabetes may be enrolled (see fasting glucose levels in inclusion criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Assessment of Change of Tumor Response Criteria in lymphoma patients During Treatment with PQR309 in patients with relapsed or refractory lymphoma according to Cheston Criteria (5) | 28 days prior to first treatment (baseline), during study treatment every 8 weeks during first 6 months and every 6 months afterwards up to 48 months
  Radiological lymphoma Evaluation (CT or other indicated according to institutional Standard practice), clinical examination and bone marrow biopsy

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs), incidence and severity of all adverse events (AEs) | During treatment on Day 1, 2, 8, 15, 22, 36 and 50; at the endof treatment and 30 days after last dose.
  Continuous and intermittent dosing
Change in pulse rate | Before treatment on Day 1,2 and after treatment started on Day 1,2, 8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in blood pressure | Before treatment on Day 1,2 and after treatment started on Day 1,2, 8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in body temperature | Before treatment on Day 1,2 and after treatment started on Day 1, 8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in ECOG (Eastern Cooperative Oncology Group) Performance Status | Before treatment on Day 1,2 and after treatment started on Day 1,8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in bodyweight/kg | Before treatment on Day 1,2 and after treatment started on Day 1,2, 8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in haematology | Before treatment on Day 1,2 and after treatment started on Day 1, 8, 15, 22, 36, 50 and subsequently every 4 weeks , at the end of treatment and 30 days after last treatment
  Continuous and intermittent dosing
Change in blood chemistry | Before treatment on Day 1and after treatment started on Day 1, 22, 50 and subsequently every 4 weeks and at the end of treatment
  Continuous and intermittent dosing
Change in haemostasis | Before treatment on Day 1and after treatment started on Day 1, 22, 50 and subsequently every 4 weeks and at the end of treatment
  Continuous and intermittent dosing
Change in ECG (electrocardiogram) | Before treatment on Day 1and after treatment started on Day 1, 22, 50 and subsequently every 4 weeks and at the end of treatment
  Continuous and intermittent dosing
Change in urine analysis | Before treatment on Day 1and after treatment started on Day 1, 22, 50 and subsequently every 4 weeks and at the end of treatment
  Continuous and intermittent dosing
Change in HbA1c | Before treatment on Day 1and after treatment started on Day 1, 22, 50 and subsequently every 4 weeks and at the end of treatment
  Continuous and intermittent dosing
Change in Cmax | During treatment on Day1, 2,8, 15,22 and 50
  Continuous and intermittent dosing
Change in tmax | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing
Change in AUC0-24 • | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing
Change in AUClast, | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing
Change in AUC0-∞, | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing
Change in t1/2 • | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing
Change in RAC • | During treatment on Day1, 2, 8, 15,22 and 50
  Continuous and intermittent dosing

OTHER OUTCOMES:
Change in insulin/ c-Peptide/ glucose | During treatment on Day 1, 2, 8,15,22 and 50
  Continuous and intermittent dosing

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, Study Director — Klinik Universität München
Locations (1):
- Medizinische Klinik und Poliklinik III, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No